CLINICAL TRIAL: NCT00895245
Title: A Phase II Clinical Trial Investigating the Efficacy of Single-Dose Fosaprepitant for the Prevention of Cisplatin-Induced Nausea and Vomiting (CINV) in Patients With Head & Neck Cancer Undergoing Concurrent Chemotherapy and Radiation
Brief Title: Fosaprepitant Dimeglumine, Palonosetron Hydrochloride, and Dexamethasone in Preventing Nausea and Vomiting Caused by Cisplatin in Patients With Stage III or Stage IV Head and Neck Cancer Undergoing Chemotherapy and Radiation Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to lack of efficacy in first 6 patients
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Keith D Eaton, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 6862; NCI-2009-01669
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-04

CONDITIONS: Nausea and Vomiting; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx
MeSH Terms: conditions — Nausea; Vomiting; Squamous Cell Carcinoma of Head and Neck | interventions — fosaprepitant; Cisplatin; Palonosetron; Dexamethasone; Calcium Dobesilate; Radiotherapy; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (Experimental): Patients receive cisplatin IV on day 1. Treatment repeats every 21 days for up to 3 courses. Patients also undergo radiotherapy once daily 5 days a week for up to 7 weeks.
  Patients receive fosaprepitant dimeglumine IV, palonosetron hydrochloride IV, and dexamethasone IV on day 1.Patients then receive oral dexamethasone on days 2-4. Patients with no emesis or requirement for rescue anti-emetics in the first 120 hours after cisplatin infusion continue to receive the anti-emetic regimen as above with the second and third courses of cisplatin.
  Patients complete an emesis diary daily for 5 days after each cisplatin infusion. Patients also complete a Functional Living Index-Emesis Questionnaire on day 8 after each cisplatin infusion.
  Interventions: Drug: fosaprepitant dimeglumine; Drug: cisplatin; Drug: palonosetron hydrochloride; Drug: dexamethasone; Other: Functional Living Index-Emesis Questionnaire; Behavioral: Emesis Diary; Radiation: Radiotherapy

INTERVENTIONS:
Drug: fosaprepitant dimeglumine — Given IV
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP; Neoplatin
Drug: palonosetron hydrochloride — Given IV
  Other Names: Aloxi; RS 25259-197
Drug: dexamethasone — Given IV and orally
  Other Names: Aeroseb-Dex; Decaderm; Decadron; Decaspray; DM; DXM
Other: Functional Living Index-Emesis Questionnaire — Ancillary studies
Behavioral: Emesis Diary — Ancillary studies
Radiation: Radiotherapy — Undergo radiotherapy
  Other Names: 3-D conformal radiotherapy or IMRT

SUMMARY:
RATIONALE: Fosaprepitant dimeglumine, palonosetron hydrochloride, and dexamethasone may help lessen or prevent nausea and vomiting caused by cisplatin in patients with head and neck cancer undergoing chemotherapy and radiation therapy.

PURPOSE: This phase II trial is studying how well fosaprepitant dimeglumine together with palonosetron hydrochloride and dexamethasone works in preventing nausea and vomiting caused by cisplatin in patients with stage III or stage IV head and neck cancer undergoing chemotherapy and radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the complete response rate of anti-emetic therapy based on a single dose of intravenous fosaprepitant with multiple cycles of high dose cisplatin (complete response is defined as no emesis or rescue nausea medications needed in the 120 hours following cisplatin infusion).

SECONDARY OBJECTIVES:

I. To determine the complete response rate of anti-emetic therapy based on a single dose of intravenous fosaprepitant with multiple cycles of high dose cisplatin in the delayed period (25-120 hours following cisplatin infusion).

II. To determine efficacy of anti-emetic therapy based on a single-dose of intravenous fosaprepitant to achieve adequate control of nausea following multiple cycles of high-dose cisplatin as defined by a score on the visual analog scale of < 25mm in the 120 hours following cisplatin infusion.

III. To determine the functional impact of cisplatin induced nausea and vomiting (CINV) on daily life as measured by the Functional Living Index-Emesis (FLIE) Questionnaire total score.

OUTLINE: Patients receive cisplatin IV on day 1. Treatment repeats every 21 days for up to 3 courses. Patients also undergo 3-D conformal radiotherapy or intensity-modulated radiotherapy once daily 5 days a week for up to 7 weeks.

Patients receive fosaprepitant dimeglumine IV, palonosetron hydrochloride IV, and dexamethasone IV on day 1 (prior to cisplatin infusion). Patients then receive oral dexamethasone on days 2-4. Patients with no emesis or requirement for rescue anti-emetics in the first 120 hours after cisplatin infusion continue to receive the anti-emetic regimen as above with the second and third courses of cisplatin.

Patients complete an emesis diary (that includes a nausea visual analog scale) daily for 5 days after each cisplatin infusion. Patients also complete a Functional Living Index-Emesis Questionnaire on day 8 of each course of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or pathologically documented squamous cell carcinoma of the oral cavity, oropharynx, larynx, hypopharynx, or nasopharynx
* Stage III or IV disease according to the AJCC Cancer Staging Handbook Sixth Edition
* Planned definitive or adjuvant radiation with concurrent cisplatin (100 mg/m2 every 3 weeks for three cycles)
* ECOG Performance Status of 0-2
* Adequate Organ Function (Hepatic: bilirubin =< 1.5 x ULN; AST and ALT =< 3 x ULN; Renal: calculated creatinine clearance >= 55ml/min (using the Cockcroft-Gault Formula); Bone Marrow: platelet count >= 100 x 10^9/L; absolute neutrophil count >= 1.25 x 10^9/L)
* Signed Informed Consent
* Male and female patients with reproductive potential must use an acceptable contraceptive method (with double barrier protection for pre-menopausal women)
* Predicted life expectancy > 12 weeks
* Willingness to complete patient diary and questionnaires

Exclusion Criteria:

* Inability or unwillingness to comply with radiotherapy or chemotherapy
* Use of illicit drugs or on-going alcohol use
* Vomiting within the 24 hours prior to cisplatin infusion
* Evidence of clinically significant congestive heart failure (Patients must be able to tolerate hydration with cisplatin)
* Peripheral Neuropathy > Grade 2
* Significant hearing loss
* Pregnant or breast-feeding women
* Patients may be enrolled in additional clinical trials, as long as no additional investigational agents are being used
* Patients with a hypersensitivity to fosaprepitant, aprepitant, polysorbate, and any other components of the EMEND product
* The following therapies are excluded during the treatment phase of the study: investigational agents; anti-neoplastic or anti-tumor agents, including immunotherapy, and hormonal anti-cancer therapy; additional scheduled anti-emetic medications, unless needed as rescue medications for acute or delayed nausea/vomiting
* Strong Inhibitors of CYP3A4: ketoconazole, itraconazole, clarithromycin, ritonavir, and nelfinavir; strong Inducers of CYP3A4: rifampin, carbamazepine, and phenytoin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-02; Primary Completion 2010-09 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Eaton, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Head and neck cancer being treated with concurrent cisplatin and radiotherapy were approached for study participation.
Groups:
- Arm I: Patients receive cisplatin IV on day 1. Treatment repeats every 21 days for up to 3 courses. Patients undergo radiotherapy once daily 5 days a week for up to 7 weeks.
  Patients receive fosaprepitant dimeglumine IV, palonosetron hydrochloride IV, and dexamethasone IV on day 1.Patients receive oral dexamethasone on days 2-4. Patients with no emesis or need for rescue anti-emetics in the first 120 hours after cisplatin continue to receive the anti-emetic regimen as above with the second and third courses of cisplatin.
  Patients complete an emesis diary daily for 5 days after each cisplatin infusion. Patients also complete a Functional Living Index-Emesis Questionnaire on day 8 after each cisplatin infusion.
  fosaprepitant dimeglumine: Given IV
  cisplatin: Given IV
  palonosetron hydrochloride: Given IV
  dexamethasone: Given IV and orally
  Functional Living Index-Emesis Questionnaire: Ancillary studies
  Emesis Diary: Ancillary studies
  Radiotherapy: Undergo radiotherapy
Period: Overall Study
Arm/Group | Arm I
Started | 6
Completed | 0
Not Completed | 6
Not completed — Lack of Efficacy | 6

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 41 [39 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With a Complete Response to the Anti-emetic Medication Regimen
Description: Complete response is defined as no emesis or rescue nausea medications needed in the first 120 hours following cisplatin infusion.
Time Frame: 120 hours following cisplatin infusion
Measure: Count of Participants; unit: Participants
Groups:
- Arm I: Patients receive cisplatin IV on day 1. Treatment repeats every 21 days for up to 3 courses. Patients undergo radiotherapy once daily 5 days a week for up to 7 weeks.
  Patients receive fosaprepitant dimeglumine IV, palonosetron hydrochloride IV, and dexamethasone IV on day 1.Patients receive oral dexamethasone on days 2-4. Patients with no emesis or need for rescue anti-emetics in the first 120 hours after cisplatin infusion continue to receive the anti-emetic regimen as above with the second and third courses of cisplatin.
  Patients complete an emesis diary daily for 5 days after each cisplatin infusion. Patients also complete a Functional Living Index-Emesis Questionnaire on day 8 after each cisplatin infusion.
  fosaprepitant dimeglumine: Given IV
  cisplatin: Given IV
  palonosetron hydrochloride: Given IV
  dexamethasone: Given IV and orally
  Functional Living Index-Emesis Questionnaire: Ancillary studies
  Emesis Diary: Ancillary studies
  Radiotherapy: Undergo r
Arm/Group | Arm I
Number analyzed (Participants) | 6
Participants | 0

2. Secondary Outcome: Rate of Complete Response to Anti-emetic Therapy in the Delayed Setting (25-120 Hours After Cisplatin Infusion)
Time Frame: 25-120 hours following cisplatin infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 6
Participants | 0

3. Secondary Outcome: Control of Nausea for 120 Hours Following Each Cisplatin Infusion for Multiple Cycles of Therapy as Measured by the Visual Analog Scale
Description: The visual analog scale ranges from 0-100. 0 is labeled as "no nausea" and 100 is labeled as "nausea as bad as it could be" A score of < 25 is considered to indicate no significant nausea. All patients discontinued trial after only one cisplatin infusion.
Time Frame: 120 hours following cisplatin infusion
Measure: Mean (Full Range); unit: millimeters
Arm/Group | Arm I
Number analyzed (Participants) | 6
millimeters | 45.2 [6 to 79]

4. Secondary Outcome: Impact of Cisplatin-induced Nausea and Vomiting on Daily Life During the 5 Day Period Following Cisplatin Infusion for Multiple Cycles as Measured by the Functional Living Index-Emesis Questionnaire
Description: FLIE is a patient-completed quality of life assessment modified from the original Functional Living Index - Cancer questionnaire. FLIE contains two domains: nausea and vomiting with nine items in each domain. The first item asks the patient to rate how much nausea (or vomiting) has occurred over a 5 day period. The remaining eight items ask patients to rate the impact of nausea (or vomiting) on various aspects of a patient's life (for example, ability to enjoy meals/liquids). Each item is answered using a 7 point visual analog scale with 7 being "none /not at all" and 1 being "a great deal". The two domains are summed for a total score with a possible range of 18-126. Higher scores indicate a more favorable quality of life. A total score of >108 defines those patients who had a minimal impact of CINV on quality of life. All particpants discontinued the trial after one cycle of cisplatin.
Time Frame: 5 days following cisplatin infusion
Population: Two patients did not complete the Functional Living Index-Emesis (FLIE) Questionnaire.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Arm I
Number analyzed (Participants) | 4
units on a scale | 83.98 [70.81 to 98.94]

ADVERSE EVENTS:
Time Frame: up to 7 weeks
Description: Only grade 2 and higher adverse events were recorded.
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=6)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Anorexia (General disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 5 (5)
leukocytes (Blood and lymphatic system disorders) | 4 (4)
Headache (Nervous system disorders) | 1 (1)
Dizziness (Ear and labyrinth disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Sinus Pain (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early due to lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes